CLINICAL TRIAL: NCT01508403
Title: A Registry Study on Shuxuetong (a Chinese Medicine Injection) Used in Twenty Hospitals
Acronym: RSCMI-I
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Collaborators: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Deputy Director, Professor, China Academy of Chinese Medical Sciences
Other Study IDs: 2009zx09502-030
Record Dates: First submitted 2011-12-20; First posted 2012-01-12 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Shuxuetong injection: a cohort using Shuxuetong injection

SUMMARY:
The purpose of this study is to make a cohort event monitoring to see whether and how Shuxuetong injection in hospital results in adverse events or adverse drug reactions.

DETAILED DESCRIPTION:
This is the first academic registry study about adverse events or adverse drug reaction for Chinese medicine injection in mainland China.

It is well known that Chinese medicine injection is just limited in mainland China, which also be accepted by China health care system.

However, more and more adverse events or adverse drug reaction have been reported in recent years in the form of case report.

In order to improving monitoring adverse events or adverse drug reaction of Chinese medicine injection in hospital, registry study will be introduced in this area.

To calculate the incidence of adverse events or adverse drug reaction is one of the main aims for this study.

According to the 'rule of three', 30,000 cases need to be registered at least.

ELIGIBILITY:
Inclusion Criteria:

* all inpatients use Shuxuetong injection in 20 selected hospitals during their hospital stay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all inpatients used or will use Shuxuetong injection in 20 selected hospitals in mainland China
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events; incidence of Shuxuetong'ADRs and identify factors that contributed to the occurrence of the adverse reaction | to assess Shuxuetong's "adverse event" and "drug adverse reaction" during patients' hospital stay, administration information of Shuxuetong will be registered every day. The registry procedure will last 3 years only for patients using Shuxuetong.
  All participants will be followed for the duration of hospital stay, an expected average of 2 weeks.Patients using Shuxuetong will be registered on a registration form including disease background, Shuxuetong's administration, and extraction information from hospital information system. An adverse event or drug adverse reaction form also will be used to describe any doubted symptoms or signs from patients. A judgment will be made by doctors directly and a further analysis will be conducted by researchers to decide those potential side effects of Shuxuetong.

CONTACTS AND LOCATIONS:
Overall Officials: Yan M Xie, Principal Investigator — Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences
Locations (1):
- Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China